CLINICAL TRIAL: NCT04519047
Title: A Randomized, Double-blind, Feasibility Study to Evaluate the Safety and Potential for Effectiveness of Intra-articular Injection of Rejoint Gel After Platelet-rich Plasma Administration in Patients With Unilateral Knee Osteoarthritis
Brief Title: IA Injection of Rejoint Gel and PRP in Patients With Unilateral Knee OA
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Collaborators: The Industrial Technology Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 201812157DSA
Record Dates: First submitted 2020-08-16; First posted 2020-08-19 (Actual); Last update posted 2020-08-24 (Actual); Status verified 2020-08

CONDITIONS: PRP; Knee Osteoarthritis
Keywords: PRP; Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Rejoint (Experimental): Rejoint+PRP
  Interventions: Biological: PRP
- Control (Active Comparator): Saline+PRP
  Interventions: Biological: PRP

INTERVENTIONS:
Biological: PRP — Beginning on treatment period, subjects will receive either Rejoint Gel or normal saline with PRP intra-articular injection twice for one month (Visit 3 and 4).

SUMMARY:
To assess the safety and tolerability of intra-articular Injection doses of Rejoint Gel after platelet-rich plasma administration in unilateral knee OA subjects.

DETAILED DESCRIPTION:
This single-center, randomized, double-blind, feasibility study to evaluate the safety and potential for effectiveness of an intraarticular Injection of Rejoint Gel after platelet-rich plasma administration in patient with single knee OA, parallel-design study will enroll approximately eligible 30 subjects with single knee OA.

The subjects will be randomized (1:1) to receive 1 of 2 treatments below:

1. Treatment Group: Rejoint Gel, intra-articular injection, with platelet-rich plasma (PRP) in 2:1 volume ratio or
2. Control Group: Normal saline, intra-articular injection with PRP in 2:1 volume ratio Beginning on treatment period, subjects will receive a single treatment cycle of either 150 mg/ml Rejoint Gel or normal saline with PRP intra-articular injection twice for one month (Visit 3 and 4). Subjects will be followed to Visit 5, 6 and 7 for safety and potential for effectiveness assessments.

ELIGIBILITY:
Inclusion criteria

1. Written informed consent before any study-specific procedure is performed;
2. Ages of 45~80 years old on the day of consent;
3. The patient is able to understand the nature of the study;
4. Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1, or 2;
5. Patient was diagnosed as OA of single knee joint by American College of Rheumatology (ACR) criteria; [i.e, knee pain, and any one of the following: age> 45 years, crepitus, or morning stiffness<30 minutes in duration, or confirmed through radiographic X ray];
6. Knee WOMAC Pain Score (sum of five components) between 20 and 40 score, after 15 meters of walking pain;
7. Contralateral knee WOMAC Pain Score <15 score;
8. Never receiving intra-articular hyaluronic acid (HA) injections of the knee, or last received intra-articular HA more than 6 months;
9. Patient meets below conditions by blood test, kidney and liver function test :

White blood cell (WBC) count > 3,000/μL Absolute neutrophil count (ANC) ≥ 1,500/μL Hemoglobin (Hb) ≥ 9.0 g/dL Thrombocyte count > 50,000/μL Blood urea nitrogen (BUN) and serum Creatinine ≤ 3X Upper Limit of Normal (ULN) Aspartate aminotransferase (AST) and Alanine aminotransferase (ALT) ≤ 3 x ULN

Exclusion criteria

1. Known sensitivity to mPEG-PLGA hydrogel (Rejoint Gel);
2. Infection in the joint or surrounding skin;
3. Known Intra-articular neoplasm;
4. Inflammatory joint disease, OA in the hips, osteonecrosis, moderate to marked effusion from index knee;
5. Documented current positive synovial fluid culture;
6. Large knee circumference (>45 cm);
7. History of herpes zoster in the past 3 months;
8. Last receiving the treatment of immunosuppressants, anti-coagulants, Non-steroidal anti-inflammatory Drugs (NSAIDs), antidepressants 14 days prior to study randomization;
9. Planned knee surgery in the next 6 months or received knee surgery in the past 6 months;
10. Subject is receiving or is less than 28 days since ending other investigational device or drug;
11. Known full-thickness cartilage loss in index knee;
12. Documented fibromyalgia, or hemiparesis;
13. Evidence of signs or symptoms of a viral, bacterial, or fungal infection occur 14 days prior to the study treatment starts, per the assessment of the investigator;
14. Any major medical or psychiatric disorder that in the opinion of the investigator, might prevent the subject from completing the study or interfere with the interpretation of the study results, such as terminal diseases, malignant tumors, heart failure (NYHA II-IV), coronary arterial disease, uncontrolled hypertension, uncontrolled diabetes, peripheral arterial disease or dementia, might prevent the subject from completing the study or interfere with the interpretation of the study results;
15. Pre-menopausal females of childbearing potential not willing to use acceptable method(s) of birth control during treatment;
16. Female subject who is lactating or pregnant

Ages: 45 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2020-08-13 (Actual); Primary Completion 2020-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Adverse events (AEs) and serious AEs | Baseline to Visit 7 (15th week)
  Adverse events (AEs) and serious AEs

SECONDARY OUTCOMES:
Western Ontario and McMaster Universities Index for osteoarthritis | Baseline to Visit 7 (15th week)
  Change in Western Ontario and McMaster Universities (WOMAC) Index for osteoarthritis: five items for pain (score range 0-20), two for stiffness (score range 0-8), and 17 for functional limitation (score range 0-68). Higher scores on the WOMAC indicate worse pain, stiffness, and functional limitations.
Kellgren-Lawrence grading scale | Baseline to Visit 7 (15th week)
  Change in the Kellgren-Lawrence (KL) Grading Scale: 0-IV (0: normal, IV: the worst)

CONTACTS AND LOCATIONS:
Overall Officials: Chueh-Hung Wu, MD, PhD, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan